CLINICAL TRIAL: NCT03163758
Title: Study of Cerebral Structural and Functional Reorganization of Stroke Patients After Repetitive Transcranial Magnetic Stimulation (rTMS) Using the Method of Neuroimaging Brain Network Analysis
Brief Title: Cerebral Reorganization of Stroke Patients After Repetitive Transcranial Magnetic Stimulation by Neuroimaging Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Chinese Academy of Sciences (Other Government); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NNSFC-81271545
Record Dates: First submitted 2017-02-20; First posted 2017-05-23 (Actual); Results first posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Stroke
Keywords: Ischemic stroke; Functional magnetic resonance imaging (fMRI); Repetitive transcranial magnetic stimulation (rTMS); Brain Reorganization
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS treatment group (Experimental): The rTMS treatment group received a 10-day real repetitive transcranial magnetic stimulation (rTMS) treatment beginning within 1 week after stroke onset.
  Interventions: Device: real Repetitive Transcranial Magnetic Stimulation
- sham group (Sham Comparator): The sham group received a 10-day sham repetitive transcranial magnetic stimulation (rTMS) treatment beginning within 1 week after stroke onset.
  Interventions: Device: sham Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: real Repetitive Transcranial Magnetic Stimulation — The rTMS treatments were performed using a Medtronic MagPro type magnetic stimulation device (Medtronic, Minneapolis, MN, USA) and a figure-of-eight coil (MC-B70, Medtronic). Coils were placed tangent to the scalp. The stimulation protocol involved 50 trains of 20 pulses applied over the ipsilesional M1 at a frequency of 5 HZ, with the stimulus intensity set at 120% of the resting motor threshold of the unaffected extremity.
  Arms: rTMS treatment group
Device: sham Repetitive Transcranial Magnetic Stimulation — The sham rTMS was performed on the same site as the rTMS treatment group but without any true stimulations. Coils were placed perpendicular to the scalp.
  Arms: sham group

SUMMARY:
The study aimed to figure out brain structural and functional reorganization evidence after repetitive transcranial magnetic stimulation through the method of neuroimaging brain network analysis, such as resting-state functional magnetic resonance imaging and diffusion tensor imaging.

ELIGIBILITY:
Inclusion Criteria:

1. stroke patients within 1 week after onset with unilateral cerebral subcortex lesion in the middle cerebral artery territory detected by diffusion weighted image,
2. right-handed,
3. without memory loss or intelligence disorder,
4. never suffered stroke before.

Exclusion Criteria:

1. direct damage to the cerebral cortex,
2. a history of cerebral vessel disease,
3. tendency to hemorrhage or existed brain hemorrhage,
4. epilepsy or other mental disorders,
5. any MRI contraindications.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-01; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li J, Zuo Z, Zhang X, Shao X, Lu J, Xue R, Fan Y, Guan Y, Zhang W. Excitatory Repetitive Transcranial Magnetic Stimulation Induces Contralesional Cortico-Cerebellar Pathways After Acute Ischemic Stroke: A Preliminary DTI Study. Front Behav Neurosci. 2018 Jul 27;12:160. doi: 10.3389/fnbeh.2018.00160. eCollection 2018. PMID 30140207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Acute ischemic stroke inpatients from the department of Neurology in Peking Union Medical College Hospital were enrolled.
Pre-assignment Details: Ten participants were excluded from the study because they didn't meet the inclusion criteria.
Period: Overall Study
Arm/Group | rTMS Treatment Group | Sham Group
Started | 21 | 21
Completed | 13 | 14
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rTMS Treatment Group | Sham Group | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (6.8) | 57.4 (14.0) | 58.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 16 | 14 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 21 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: National Institutes of Health Stroke Scale (NIHSS)
Description: The investigators use National Institutes of Health Stroke Scale (NIHSS) to evaluate the participants' neural deficit after stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0. Higher NIHSS scores mean a worse outcome.
Time Frame: Change from Baseline NIHSS at 1 month after real rTMS/sham rTMS
Population: Two patients lost in the follow-up of the rTMS treatment group. And three patients lost in the follow-up of the sham group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS Treatment Group | Sham Group
Number analyzed (Participants) | 19 | 18
score on a scale | 3.8 (1.8) | 2.7 (0.6)

2. Primary Outcome: Barthel Index (BI)
Description: The investigators use Barthel Index (BI) to evaluate the participants' activities of daily living after stroke. The BI consists of 10 questions that relate to degree of independence with activities of daily living, including toileting, bathing, eating, dressing, continence, transfers, and ambulation. The BI score is calculated by summing the response value to each of the 10 questions. The BI score ranges from 0 to 100. A patient scoring 0 points would be dependent in all assessed activities of daily living, whereas a score of 100 would reflect independence in these activities. A higher score is associated with a better outcome.
Time Frame: Change from Baseline BI at 1 month after real rTMS/sham rTMS
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS Treatment Group | Sham Group
Number analyzed (Participants) | 19 | 18
score on a scale | 22.6 (6.5) | 17.8 (6.9)

3. Primary Outcome: Fugl-Meyer Assessment Upper Limb (FMA-UL)
Description: The investigators use Fugl-Meyer assessment Upper Limb (FMA-UL) to evaluate the participants' motor function of upper limb. The FMA-UL is an ordinal scale that has 3 points for each item. A zero score is given for the item if the subject cannot do the task. A score of 1 is given when the task is performed partially and a score of 2 is given when the task is performed fully. The maximum score of FMA-UL is 66 and the minimum score is 0. Higher scores mean a better outcome.
Time Frame: Change from Baseline FMA at 1 month after real rTMS/sham rTMS
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS Treatment Group | Sham Group
Number analyzed (Participants) | 19 | 18
score on a scale | 14.9 (4.4) | 11.1 (3.8)

4. Secondary Outcome: Functional Connectivity Map (FC Map)
Description: Functional Connectivity was examined using a seed-based voxel-wise correlation approach. The ipsilesional primary motor cortex (M1) was defined as the region of interest. Pearson's correlation analysis between the time course of the ipsilesional M1 and that of every voxel in the whole brain was computed for a map of correlation coefficients, which were Fisher's z-transformed and called as z-FC maps.
Time Frame: Change from Baseline z-FC maps at 1 month after real rTMS/sham rTMS
Population: This outcome measurement, the z-FC map, is not numeric data. Z-FC map is a radiographic imaging measurement. The study compared the difference of the z-FC map between the rTMS treatment group and the sham group.
Arm/Group | rTMS Treatment Group | Sham Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: one month after real/sham rTMS treatment
Description: The common adverse events of rTMS are headache, dizzy, scalp discomfort at the site of stimulation, tingling, spasms or twitching of facial muscles and lightheadedness. The uncommon side effects of rTMS include seizures, mania, and hearing loss.
Arm/Group | rTMS Treatment Group | Sham Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 2/21 | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rTMS Treatment Group (N=21) | Sham Group (N=21)
headache (Nervous system disorders) | 1 (1) | 1 (1)
dizzy (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-01-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT03163758/Prot_SAP_000.pdf